CLINICAL TRIAL: NCT06276907
Title: An Open-label Randomized Controlled Trial Comparing the Role of Therapeutic Plasma-exchange in Ameliorating Secondary Organ Dysfunctions in Patients With ACLF and Develop Biomarkers of Treatment Response
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-16
Record Dates: First submitted 2024-01-02; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma Exchange (Experimental): On day 1 Response assessment will be done to assess the need for a second session from day 3-7 and subsequently every week till day 28. A minimum of 3 sessions would be considered in the first seven days. The duration of each session would be 3-4 hours. Patients with partial response (not meeting criteria for a complete response after 3 sessions) would be considered for additional sessions as decided by the treating physician until desired complete response, adverse effects, liver transplant, death, or clinical futility. The complete response will be defined as a sustained reduction in bilirubin and international normalized ratio without any clinical worsening requiring discontinuation of therapy. Failure of therapy would be defined as the development of adverse effects, new onset sepsis, or organ failure. In such patients, further sessions would be deferred. Blood access was established with a double-lumen catheter inserted into the patient's femoral or jugular vein.
  Interventions: Biological: Plasma Exchange
- Standard Medical Treatment (Active Comparator): Patients randomized to SMT Group will be given standard medical therapy (SMT) only included as per requirement.
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: Plasma Exchange — On day 1 Response assessment will be done to assess the need for a second session from day 3-7 and subsequently every week till day 28. A minimum of 3 sessions would be considered in the first seven days. The duration of each session would be 3-4 hours. Patients with partial response (not meeting criteria for a complete response after 3 sessions) would be considered for additional sessions as decided by the treating physician until desired complete response, adverse effects, liver transplant, death, or clinical futility. The complete response will be defined as a sustained reduction in bilirubin and international normalized ratio without any clinical worsening requiring discontinuation of therapy. Failure of therapy would be defined as the development of adverse effects, new onset sepsis, or organ failure. In such patients, further sessions would be deferred. Blood access was established with a double-lumen catheter inserted into the patient's femoral or jugular vein.
  Arms: Plasma Exchange
Other: Standard Medical Treatment — Patients randomized to SMT Group will be given standard medical therapy (SMT) only included as per requirement.
  Arms: Standard Medical Treatment

SUMMARY:
Rationale: Current understanding of the pathophysiology of ACLF suggests that unresolved injury, poor infection control, and liver regeneration result in persistent systemic inflammation and cytokine storm, which subsequently lead to systemic inflammatory response syndrome (SIRS) resulting in multiple organ failures, septic shock and deaths in ACLF. Nearly 74% of ACLF patients initially diagnosed without SIRS, sepsis, or organ failure developed SIRS by day 7 which increases the onset of secondary organ failure and sepsis with high short-term mortality. The emerging use of plasma exchange has shown some potential benefits in terms of dampening systemic inflammation and improvement of outcomes in some ACLF patients. However, there is currently no randomized controlled trial exploring the potential role in ameliorating secondary organ dysfunctions in patients with ACLF is not known. Hence in the current objective, we want to study the role of plasma exchange in the management of sec. organ failure in ACLF patients in a randomized controlled trial and identify the biomarker to access the treatment response to therapy.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that detrimental complications which include secondary organ dysfunction (circulation, brain, respiration, and kidneys) in patients with acute on chronic liver failure may be related to defects in the host response, which may be responsible for the progression of the disease. Thus, understanding the pathophysiology of secondary organ dysfunction particularly the role of gut dysbiosis and metabolic adaptation of the host in patients with ACLF is essential for preventing and ameliorating the function of these organs which in turn would improve overall survival. Considering systemic inflammation induces metabolic adaptation, the role of TPE in preventing the development of secondary organ failures and biomarkers of response to therapy would be evaluated in patients with ACLF.

Key Objectives: Can we develop specific biomarkers of response to therapy to identify the right patient selection that could benefit from spontaneous survival and avoid a liver transplant? Primary Objective To study the role of therapeutic plasma exchange versus standard medical treatment in patients with ACLF on improving AARC grade by 1 at day 14.

Secondary Objectives

* To study the role of TPE versus standard medical treatment in patients with ACLF on transplant-free survival at 28-days
* To study the impact on progression or resolution of secondary organ failures at day 7 and 14
* Impact on systemic inflammation, renal functions, and ammonia at day 3 7, and day 14
* Impact on systemic hemodynamics- decrease in the dose of vasopressors, lactate clearance, and improvement in PaO2/FiO2 ratio and urine output after therapy
* Impact on bilirubin and bile acid reduction at day 3 7 and 14
* Impact on the development of infections, new organ failures at day 7 and day 14
* To study the levels of CRP, IL-6, IL-10 pre and post-therapy at day 3, 7 and 14
* To evaluate the improvement in AARC, SOFA and MELD at day 3 7, 14 and develop a model based on AARC score for identifying responders.
* Adverse effects of therapy
* Additional experiments of plasma proteomics and metabolomics will be performed. (as mentioned above)
* To study the impact on systemic inflammation, endothelial function (von-willebrand factor and ADAMTS), inflammatory cytokines damage-associated molecular patterns (HMGB1) at day 3 and 7 and day 14
* Impact on monocyte function (phagocytosis and mitochondrial respiration) In this open-label, randomized controlled trial patients will be randomized 1:1 to two groups. Patients would be randomized using block randomization with 19 blocks and block-size of 10 and SNOSE technique (sequentially numbered opaque sealed envelopes). Patients fulfilling the selection criteria of ACLF AARC consensus will be recruited in the study and will be randomized into two groups patients in each group) to receive either standard medical therapy alone or standard therapy with plasma-exchange (details mentioned below).

Interventions SMT Group: Patients randomized to SMT Group will be given standard medical therapy (SMT) only included as per requirement. Nutritional therapy 25-30 kcal/kg/day, to reach at least 80% of this target, lactulose, bowel wash, albumin, terlipressin or norepinephrine, and antibiotics will be provided according to the local institutional guidelines. Anti-virals in hepatitis B reactivation and details of the type of antiviral will be included..

Patients with organ failures requiring organ support would be managed in the intensive care unit. Patients would be managed with the standard of care which will include the use of vasopressors (norepinephrine or terlipressin for maintaining mean arterial pressure >65 mm of Hg, non-invasive or invasive mechanical ventilation, renal replacement therapy ( intermittent or continuous renal replacement therapy) for standard renal indications. Patients would be fed enterally with the use of parenteral nutrition in patients wherein enteral nutrition is not tolerated. Intravenous low-dose hydrocortisone would be administered to patients with norepinephrine >0.25 ug/kg/min, according to Surviving Sepsis Campaign Guidelines 2021. The use of antioxidants (N-acetylcysteine) would be recorded.

Plasma exchange: Patients randomized to this group will receive plasma exchange on day 1 Response assessment will be done to assess the need for a second session from day 3-7 and subsequently every week till day 28. A minimum of 3 sessions would be considered in the first seven days. The duration of each session would be 3-4 hours. Patients with partial response (not meeting criteria for a complete response after 3 sessions) would be considered for additional sessions as decided by the treating physician until desired complete response, adverse effects, liver transplant, death, or clinical futility. The complete response will be defined as a sustained reduction in bilirubin and international normalized ratio without any clinical worsening requiring discontinuation of therapy. Failure of therapy would be defined as the development of adverse eff ects, new onset sepsis, or organ failure. In such patients, further sessions would be deferred. Blood access was established with a double-lumen catheter inserted into the patient's femoral or jugular vein.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ACLF with AARC grade 2 or more with or without single secondary organ failure.

Exclusion Criteria:

1. 1. Patients with age less than 18 years or more than 65 years
2. Patients with HVOTO or EHPVO
3. Hepatocellular carcinoma (beyond Milan) or any extrahepatic malignancy
4. Active bleed (mucosal or variceal) or severe coagulopathy (platelets <20,000 or INR>4)
5. Patients with refractory shock requiring norepinephrine >0.5ug/kg/min
6. Patients with retroviral infections
7. Pregnancy or active breastfeeding
8. Known severe cardiopulmonary diseases (structural or valvular heart disease, coronary artery disease, coronary pulmonary disease, chronic kidney disease)
9. Lack of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The AARC grading is done by AARC score the values of which vary from 5-15 , pts are divided into 3 grades i.e AARC score 5-7- grade 1, 8-10- grade 2, and AARC 11-15 as grade 3. Improvement in 1 grade is associated with 40% improvement in 28-day survival | 28 days
  the measure is an ordinal variable with 3 categories as above (grade 1, 2 and 3) derived from AARC score from 5-15

SECONDARY OUTCOMES:
Transplant-free survival at 28-days | 28 days
The impact of TPE on the progression or resolution of secondary organ failures at day 7, 14 and 28 | day 7, 14 and 28
  Each organ failure will be defined based on the definition as yes or no. Depending on if the patient improves or progresses the information will be collected and analyzed.
the development of infection at day 7 and 14 in patients who had no infection | day 7 and day 14
Duration of ICU and hospital stay | 28 days
The proportion of patients developing adverse events will be compared between the two groups | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided